CLINICAL TRIAL: NCT06656546
Title: Comparison of Three Ultrasound Methods for Assessment of Endotracheal Tube Placement During Intubation: A Randomised Study
Brief Title: Comparison of Ultrasound Methods for Assessment of Endotracheal Tube Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emre Kudu, Principal Investigator, Marmara University Pendik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 09.2024.629
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Intubation; Difficult or Failed
Keywords: Ultrasonography; Rapid sequence intubation; End-tidal carbondioxide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: During the endotracheal intubation procedure, the intubation itself and associated interventions will be performed by the patient's attending physician and healthcare team. The ultrasound operator, who will be blinded to the intubation process and its outcomes, will wear soundproof headphones to ensure no external auditory cues influence their assessment. The ultrasound operator will determine the intubation placement solely based on their ultrasound findings, and only the operator will have access to the ultrasound images. The rest of the team will remain blinded to the ultrasound results. Additionally, a designated individual will record the duration of the procedures for both the intubation and ultrasound teams to ensure accurate time tracking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tracheal Ultrasound (Experimental): The success of endotracheal intubation (ETI) will be checked by tracheal ultrasonography. The primary outcome will be the placement of the endotracheal tube (ETT) in the trachea or esophagus. The secondary outcome will assess the duration of the ultrasound procedure. The time measurement will begin immediately after the placement of the ETT and will continue until a decision is made, via ultrasound, regarding whether the intubation is tracheal or esophageal.
  Interventions: Diagnostic Test: Tracheal Ultrasound
- Lung Ultrasound (Experimental): The success of ETI will be checked by lung ultrasonography. The primary outcome will be the placement of the ETT in the trachea or esophagus. The secondary outcome will assess endobronchial intubation and the duration of the ultrasound procedure. The time measurement will begin immediately after the placement of the ETT and will continue until a decision is made, via ultrasound, regarding whether the intubation is tracheal or esophageal.
  Interventions: Diagnostic Test: Lung Ultrasound
- Diaphragm Ultrasound (Experimental): The success of ETI will be checked by diaphragm ultrasonography. The primary outcome will be the placement of the ETT in the trachea or esophagus. The secondary outcome will assess endobronchial intubation and the duration of the ultrasound procedure. The time measurement will begin immediately after the placement of the ETT and will continue until a decision is made, via ultrasound, regarding whether the intubation is tracheal or esophageal.
  Interventions: Diagnostic Test: Diaphragm Ultrasound

INTERVENTIONS:
Diagnostic Test: Tracheal Ultrasound — In the clinic, one of the routinely used ultrasound machines, either the HM70 EVO Linear Probe (5-12 MHz) or the eSaote MyLab Seven Linear Probe (3-13 MHz), will be selected based on suitability for the procedure at the time. A linear transducer will be placed perpendicular to the trachea at the level of the cricoid membrane. During ETI, visualization of the ETT moving within the trachea, specifically behind the cricothyroid membrane, indicates successful intubation. In contrast, if the ETT is mistakenly placed in the esophagus, a double-lumen appearance lateral to the trachea, created by the ETT within the esophagus, suggests esophageal intubation.
  Arms: Tracheal Ultrasound
Diagnostic Test: Lung Ultrasound — In the clinic, one of the routinely used ultrasound machines, either the HM70 EVO Linear Probe (5-12 MHz) or the eSaote MyLab Seven Linear Probe (3-13 MHz), will be selected based on suitability for the procedure at the time. Following ETI, the presence of lung sliding will be evaluated using ultrasound with the aid of a linear probe.The transducer will be placed bilaterally along the mid-axillary line, between the second and fifth intercostal spaces, in a coronal orientation. After the ETT is placed and ventilation is initiated, the movement of the visceral and parietal pleura will be assessed. The presence of sliding motion between these pleural layers during ventilation indicates successful intubation, whereas the absence of this movement suggests a failed intubation.
  Other Names: Lung Sliding
  Arms: Lung Ultrasound
Diagnostic Test: Diaphragm Ultrasound — In the clinic, one of the routinely used ultrasound machines, either the HM70 EVO Curvilinear Probe (2-8 MHz) or the eSaote MyLab Seven Curvilinear Probe (1-8 MHz), will be selected based on suitability for the procedure at the time. Using a curvilinear transducer, the probe will be placed along the mid-axillary line, approximately at the seventh to ninth intercostal spaces, in a coronal orientation. The movement of the diaphragm during ventilation will be assessed over the spleen and liver. Diaphragmatic motion during ventilation indicates successful ETI, while the absence of bilateral diaphragmatic movement suggests esophageal intubation. If diaphragmatic movement is only observed on one side, it is indicative of endobronchial intubation.
  Other Names: Diaphragm Excursion
  Arms: Diaphragm Ultrasound

SUMMARY:
This study is a single-center, randomized clinical trial conducted in an emergency department on intubated patients with rapid sequence intubation. Two sonographers will independently verify the accuracy of the intubation site using the assigned intubation method (tracheal, lung-sliding, or diaphragm) according to the randomization sequence. Each sonographer will be blinded to the other verification methods (physical examination, end-tidal carbon dioxide) being used. The study's primary objective is to compare the diagnostic accuracy of different intubation techniques.

DETAILED DESCRIPTION:
In emergency medicine, endotracheal intubation (ETI) is commonly performed for patients who require airway management due to acute respiratory failure, inadequate oxygenation or ventilation, or an inability to protect the airway resulting from altered consciousness. When ETI is performed outside of a cardiac arrest scenario, a series of steps are followed to optimize the procedure. These steps aim to prevent hypoxia, maintain hemodynamic stability, reduce the risk of aspiration, and increase the success rate of ETI. This methodical approach is known as Rapid Sequence Intubation (RSI). RSI involves preparing the necessary and auxiliary equipment, administering premedication, ensuring oxygenation, and applying anesthetic and neuromuscular blocking agents, followed by the placement of the endotracheal tube (ETT). The procedure concludes with confirming the ETT's placement and providing post-intubation care.

The primary goal of ETI is to position the ETT through the vocal cords into the trachea, ensuring that both lungs are ventilated effectively. Incorrect or unrecognized endobronchial intubation can result in hypoventilation and collapse of the non-ventilated lung, while the over-ventilated lung may suffer barotrauma or pneumothorax. Unrecognized esophageal intubation, on the other hand, can lead to failure in ventilation, resulting in hypoxia and subsequent complications, including brain damage and other morbidities. Therefore, ensuring the correct placement of the ETT is crucial to avoid serious adverse outcomes.

Various methods have been described to confirm correct ETT placement, including direct visualization during intubation, observation of chest wall movements, bilateral auscultation of lung sounds, end-tidal carbon dioxide (EtCO2) monitoring, fiberoptic bronchoscopy, and chest X-ray. Among these, capnography is considered the gold standard. However, in specific clinical situations, EtCO2 monitoring may be unreliable. Patients in cardiac arrest, patients with severe hypotension, pulmonary embolism, or poor pulmonary reserve may present lower than expected EtCO2 values. Similarly, gastric insufflation, using antacids, or consuming carbonated beverages may result in false-positive readings.

The American College of Emergency Physicians (ACEP) guidelines recommend the use of additional confirmation methods after ETT placement. Ultrasound (US) has emerged as a relatively new technique for confirming ETI. Its advantages include being non-invasive, portable, rapid, and capable of providing real-time, accurate results. Additionally, the US is unaffected by environmental noise, which can be challenging in noisy environments such as the emergency department. It is also not influenced by changes in pulmonary blood flow.

Several ultrasound techniques have been described to confirm ETT placement. The most commonly used methods include direct visualization of the ETT during intubation (tracheal ultrasound), detection of the "lung sliding" sign via lung ultrasound to indicate lung aeration and bilateral identification of diaphragmatic movement. Tracheal ultrasound can detect esophageal intubation before ventilation begins, preventing unnecessary gastric insufflation and its associated complications. The lung sliding sign and bilateral diaphragmatic movement techniques can help identify endobronchial intubation by visualizing pleural and diaphragmatic movement, respectively, thereby complementing tracheal ultrasound and reducing the risk of missed endobronchial intubation.

A comprehensive literature review revealed that no studies have directly compared these three ultrasound methods. Therefore, this study aims to evaluate the effectiveness of these three ultrasound techniques in confirming ETT placement and to compare the time required for each method. A secondary objective is to compare the time spent using ultrasound with that of auscultation and capnography. Additionally, this study will assess the ability of each ultrasound technique to detect tracheal intubation and, if present, accidental esophageal intubation across all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the emergency department who require endotracheal intubation (ETI) based on the decision of the primary physician and are intubated using the rapid sequence intubation method.
* Patients aged >18 years will be included in the study.

Exclusion Criteria:

* Pregnant patients.
* Patients with a history of neck or chest surgery that may interfere with ultrasound evaluation.
* Patients with cervical spine disease or a history of surgery that could affect diaphragmatic movement.
* Patients diagnosed conditions such as pneumothorax that could affect lung ultrasound results, or those in whom pneumothorax is detected upon further evaluation,
* Patients who, after being enrolled, withdraw consent either personally or through a relative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Endotracheal Intubation Success | Immediately after intubation, assessed within the first 5 minutes after the procedure.
  The primary outcome is the success of endotracheal intubation. The decision will be made by the primary physician based on routine clinical practice and current guidelines. Physical examination and end-tidal carbon dioxide monitoring will be used, among other methods, to assist in this decision. The primary physician will determine at the bedside whether the intubation was successful (tracheal intubation) or unsuccessful (esophageal intubation). Neither the ultrasound operator nor anyone else will intervene in the decision-making process.

SECONDARY OUTCOMES:
Endotracheal Intubation Confirmation Time | Immediately after intubation, assessed within the first 5 minutes after the procedure.
  The duration of each method used to confirm endotracheal intubation (ultrasonography, physical examination, and end-tidal carbon dioxide) will be recorded separately. The timing will start from the placement of the endotracheal tube and connection to the bag-valve mask, and will end once a determination-successful (tracheal intubation) or unsuccessful (esophageal intubation)-is made using the respective method. If the primary physician determines esophageal intubation, the remaining uncompleted methods will be discontinued to avoid disrupting the patient's routine management or causing harm. If the ultrasonography procedure is not completed, it will be considered unsuccessful.
  The timing will begin after the completion of intubation and connection to the bag-valve mask, and will continue until a decision is made. The total duration will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Kudu, MD, Study Director — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acquisto NM, Mosier JM, Bittner EA, Patanwala AE, Hirsch KG, Hargwood P, Oropello JM, Bodkin RP, Groth CM, Kaucher KA, Slampak-Cindric AA, Manno EM, Mayer SA, Peterson LN, Fulmer J, Galton C, Bleck TP, Chase K, Heffner AC, Gunnerson KJ, Boling B, Murray MJ. Society of Critical Care Medicine Clinical Practice Guidelines for Rapid Sequence Intubation in the Critically Ill Adult Patient. Crit Care Med. 2023 Oct 1;51(10):1411-1430. doi: 10.1097/CCM.0000000000006000. Epub 2023 Sep 14. PMID 37707379
- [Background] Drescher MJ, Conard FU, Schamban NE. Identification and description of esophageal intubation using ultrasound. Acad Emerg Med. 2000 Jun;7(6):722-5. doi: 10.1111/j.1553-2712.2000.tb02055.x. No abstract available. PMID 10905655
- [Background] Roy PS, Joshi N, Garg M, Meena R, Bhati S. Comparison of ultrasonography, clinical method and capnography for detecting correct endotracheal tube placement- A prospective, observational study. Indian J Anaesth. 2022 Dec;66(12):826-831. doi: 10.4103/ija.ija_240_22. Epub 2022 Dec 20. PMID 36654895
- [Background] Chou HC, Tseng WP, Wang CH, Ma MH, Wang HP, Huang PC, Sim SS, Liao YC, Chen SY, Hsu CY, Yen ZS, Chang WT, Huang CH, Lien WC, Chen SC. Tracheal rapid ultrasound exam (T.R.U.E.) for confirming endotracheal tube placement during emergency intubation. Resuscitation. 2011 Oct;82(10):1279-84. doi: 10.1016/j.resuscitation.2011.05.016. Epub 2011 Jun 1. PMID 21684668
- [Background] Sethi AK, Salhotra R, Chandra M, Mohta M, Bhatt S, Kayina CA. Confirmation of placement of endotracheal tube - A comparative observational pilot study of three ultrasound methods. J Anaesthesiol Clin Pharmacol. 2019 Jul-Sep;35(3):353-358. doi: 10.4103/joacp.JOACP_317_18. PMID 31543584
- [Background] Werner SL, Smith CE, Goldstein JR, Jones RA, Cydulka RK. Pilot study to evaluate the accuracy of ultrasonography in confirming endotracheal tube placement. Ann Emerg Med. 2007 Jan;49(1):75-80. doi: 10.1016/j.annemergmed.2006.07.004. Epub 2006 Oct 2. PMID 17014927
- [Background] Lin J, Bellinger R, Shedd A, Wolfshohl J, Walker J, Healy J, Taylor J, Chao K, Yen YH, Tzeng CT, Chou EH. Point-of-Care Ultrasound in Airway Evaluation and Management: A Comprehensive Review. Diagnostics (Basel). 2023 Apr 25;13(9):1541. doi: 10.3390/diagnostics13091541. PMID 37174933